CLINICAL TRIAL: NCT05976152
Title: Effect of Butyphthalide on Cognitive Level Change After Cerebral Vascular Event-a Randomized Control Trial (Be-CLEVER)
Acronym: Be-CLEVER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Qiang Dong, Director of Neurology Department, Huashan Hospital, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Be-CLEVER
Record Dates: First submitted 2023-07-06; First posted 2023-08-04 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Post-stroke Cognitive Impairment (PSCI)
Keywords: stroke; PSCI; Butylphthalide
MeSH Terms: conditions — Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dl-3-butylphthalide (Experimental): Routine treatment and dl-3-butylphthalide
  Interventions: Drug: dl-3-butylphthalide; Drug: dl-3-butylphthalide placebo
- dl-3-butylphthalide Placebo (Placebo Comparator): Routine treatment and dl-3-butylphthalide Placebo
  Interventions: Drug: dl-3-butylphthalide; Drug: dl-3-butylphthalide placebo

INTERVENTIONS:
Drug: dl-3-butylphthalide — First stage： Routine stroke treatment: hypoglycemic, antihypertensive, antiplatelet, anticoagulant and other conventional cerebrovascular disease treatment drugs.
  Placebo group: routine stroke treatment + oral Butylphthalide Placebo Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Butylphthalide group: routine stroke treatment + oral Butylphthalide Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Second stage： 14d washout period after first stage. Routine PSCI treatment: 5-10 mg Donepezil, qd. Placebo group: Routine PSCI treatment + oral Butylphthalide Placebo Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Butylphthalide group:
  Routine PSCI treatment + oral Butylphthalide Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Other Names: DL-3-n-butylphthalide (NBP)
Drug: dl-3-butylphthalide placebo — First stage： Routine stroke treatment: hypoglycemic, antihypertensive, antiplatelet, anticoagulant and other conventional cerebrovascular disease treatment drugs.
  Placebo group: routine stroke treatment + oral Butylphthalide Placebo Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Butylphthalide group: routine stroke treatment + oral Butylphthalide Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Second stage： 14d washout period after first stage. Routine PSCI treatment: 5-10 mg Donepezil, qd. Placebo group: Routine PSCI treatment + oral Butylphthalide Placebo Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Butylphthalide group:
  Routine PSCI treatment + oral Butylphthalide Soft Capsules, 2 capsules/time, tid, an empty stomach for 24 weeks.
  Other Names: NBP placebo

SUMMARY:
Post-stroke cognitive impairment (PSCI) refers to a clinical syndrome characterized by cognitive impairment that occurs after a stroke event and persists for at least 24 weeks. Due to the early recovery of conditions such as delirium and transient cognitive impairment after stroke, the diagnosis of PSCI often requires cognitive assessment at 12 to 24 weeks post-stroke to determine the severity of cognitive impairment. It can be classified according to the severity of cognitive impairment as post-stroke cognitive impairment no dementia (PSCIND) and post-stroke dementia (PSD). Recent large international cohort studies have reported an incidence rate of PSCI ranging from 24% to 53.4%, and patients with PSCI have a significantly higher mortality rate compared to those without cognitive impairment. Guidelines such as American Heart Association/American Society of Anesthesiologists (AHA/ASA) and the Chinese "Expert Consensus on the Management of Post-Stroke Cognitive Impairment" propose integrating cognitive impairment and stroke intervention strategies. Early comprehensive intervention and treatment for high-risk individuals after stroke, aiming to delay or prevent the progression from PSCIND to PSD, are the primary goals in the current treatment of PSCI. However, there is currently a lack of large randomized controlled trials (RCTs) for PSCI, and research is still needed to determine whether cognitive-enhancing drugs can reduce the risk of PSCI occurrence and improve outcomes and prognosis for PSCI patients. A randomized, double-blind, multicenter clinical study involving 281 non-dementia vascular cognitive impairment (VCI) patients showed that the overall cognitive scores of patients treated with donepezil for 24 weeks significantly improved compared to the placebo group.

The aim of this study is to evaluate the effectiveness of donepezil in the treatment of post-stroke cognitive impairment. It will be a multicenter, randomized, double-blind, placebo-controlled trial with a 48-week treatment duration. The study will observe the difference in PSCI incidence rate between the donepezil treatment group and the conventional stroke treatment group at 24 weeks and evaluate the improvement in post-stroke cognitive impairment after 6 months of donepezil treatment compared to conventional treatment.

This study will be conducted in two stages: the first stage (0-24 weeks) aims to assess whether donepezil can reduce the risk of PSCI occurrence and will be a multicenter, randomized, double-blind, placebo-controlled study. The second stage (24-48 weeks) aims to evaluate whether donepezil can improve the prognosis of PSCI patients and will also be a multicenter, randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

First stage:

* Acute ischemic stroke (AIS) symptom onset within 14 days Signs and symptoms consistent with the diagnosis of an acute ischemic stroke by CT/MRI.
* Age >= 60 years，
* Baseline NIHSS 3-18.
* Patient can complete questionnaire survey, physical examination, cranial MRI and other medical examinations
* Patient/legally authorized representative has signed the Informed Consent Form

Second stage:

* Patient with stage I diagnosis of PSCI.
* Patient can complete questionnaire survey, physical examination, cranial MRI and other medical examinations.
* Patient/legally authorized representative has signed the Informed Consent Form

Exclusion Criteria:

First stage:

* Patients who had been diagnosed with dementia prior to stroke
* Other related factors affecting cognitive function: central nervous system infection, neurodegenerative diseases, trauma, poisoning, intracranial space occupying lesions, metabolic diseases, etc.
* Other serious central nervous system diseases: Parkinson's disease, epilepsy, multiple sclerosis, motor neurone disease, immune-related encephalomyelopathy, etc.
* Serious mental illness: anxiety disorder, depression, delirium, schizophrenia, bipolar disorder, mental retardation, which is diagnosed or controlled by medication.
* Uncorrectable visual and hearing impairments and inability to complete neuropsychological tests
* Severe liver and kidney dysfunction
* The presence of a malignant tumor or other serious/life-threatening disease that could cause the subject's death within 12 months.
* Current known alcohol or illicit drug abuse or dependence
* Patients undergoing thrombectomy, thrombolysis, carotid endarterectomy, or other surgical procedures during the acute infarction.
* Using cholinesterase inhibitors, N-methyl-D-aspartate (NMDA) receptor antagonists, or Sodium oligomannate (GV-971).
* Allergic to any component of butylphthalein
* Pregnancy or lactation, have the possibility of becoming pregnant, and who plan to become pregnant
* Participants in other interventional clinical trials
* MRI contraindications (e.g., claustrophobia, hypersensitivity to contrast media, etc.)

Second stage:

* During the first phase of follow-up, participants' compliance was poor, with study medication compliance less than 80% or greater than 120%; Follow-up was less than 24 weeks or did not complete the follow-up within the follow-up window..
* Recurrent stroke in the first stage

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PSCI incidence | 24 weeks (first stage)
  Compared with routine stroke treatment, the difference of the PSCI incidence at 24 weeks with butylphthalide treatment.
vadas-cog score | 6 months (Second stage)
  Compared with routine treatment, improvement of vadas-cog scores at 24 weeks with butylphthalide treatment

SECONDARY OUTCOMES:
Changes of Montreal Cognitive Assessment (MoCA) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Montreal Cognitive Assessment (MoCA) at 24 weeks compared with baseline
Changes of Mini-Mental State Examination (MMSE) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Mini-Mental State Examination (MMSE) at 24 weeks compared with baseline
Changes of Neuropsychiatric Inventory Questionnaire (NPI-Q) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Neuropsychiatric Inventory Questionnaire (NPI-Q) at 24 weeks compared with baseline
Changes of Hamilton Anxiety Scale (HAMA) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Hamilton Anxiety Scale (HAMA) at 24 weeks compared with baseline
Changes of Hamilton Depression Scale (HAMD) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Hamilton Depression Scale (HAMD) at 24 weeks compared with baseline
Changes of 23-item version of Alzheimer's Disease Cooperative Study- activities of daily living scale (ADCS-ADL23) for activities of daily living at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of 23-item version of Alzheimer's Disease Cooperative Study- activities of daily living scale (ADCS-ADL23) for activities of daily living at 24 weeks compared with baseline
Changes of Clinical Dementia Rating (CDR) at 24 weeks compared with baseline | 24 weeks (first stage)
  Changes of Clinical Dementia Rating (CDR) at 24 weeks compared with baseline
Changes of infarct volume by cranial magnetic resonance imaging (MRI) at 24 weeks after treatment with butylphthalein compared with routine stroke treatment. | 24 weeks (first stage)
  Changes of infarct volume by cranial magnetic resonance imaging (MRI) at 24 weeks after treatment with butylphthalein compared with routine stroke treatment.
Changes of infarct location by cranial magnetic resonance imaging (MRI) at 24 weeks after treatment with butylphthalein compared with routine stroke treatment. | 24 weeks (first stage)
  Changes of infarct location by cranial magnetic resonance imaging (MRI) at 24 weeks after treatment with butylphthalein compared with routine stroke treatment.
stroke recurrence | 24 weeks (first stage)
  Difference in stroke recurrence rate of butylphthalein treatment compared with routine stroke treatment at 24 weeks
Changes of modified Rankin Scale score (mRS) at 24 weeks compared with baseline. | 24 weeks (first stage)
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The mRS is a range from 0-6. 0=No symptoms, 1=No significant disability. Able to carry out all usual activities, despite some symptoms. 2=Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3=Moderate disability. Requires some help, but able to walk unassisted. 4=Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5=Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6=Dead
Changes of Montreal Cognitive Assessment (MoCA) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Montreal Cognitive Assessment (MoCA) at 48 weeks compared with baseline
Changes of Mini-Mental State Examination (MMSE) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Mini-Mental State Examination (MMSE) at 48 weeks compared with baseline
Changes cognitive domain level by Symbol Digit Modalities Test at 48 weeks compared with baselinel | 48 weeks (second stage)
  Changes cognitive domain level by Symbol Digit Modalities Test at 48 weeks compared with baseline
Changes cognitive domain level by Trail Making Test at 48 weeks compared with baseline. | 48 weeks (second stage)
  Changes cognitive domain level by Trail Making Test at 48 weeks compared with baseline.
Changes of Neuropsychiatric Inventory Questionnaire (NPI-Q) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Neuropsychiatric Inventory Questionnaire (NPI-Q) at 48 weeks compared with baseline
Changes of Hamilton Anxiety Scale (HAMA) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Hamilton Anxiety Scale (HAMA) at 48 weeks compared with baseline
Changes of Hamilton Depression Scale (HAMD) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Hamilton Depression Scale (HAMD) at 48 weeks compared with baseline
Changes of Clinical Dementia Rating (CDR) at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of Clinical Dementia Rating (CDR) at 48 weeks compared with baseline
Changes of 23-item version of Alzheimer's Disease Cooperative Study- activities of daily living scale (ADCS-ADL23) for activities of daily living at 48 weeks compared with baseline | 48 weeks (second stage)
  Changes of 23-item version of Alzheimer's Disease Cooperative Study- activities of daily living scale (ADCS-ADL23) for activities of daily living at 48 weeks compared with baseline
stroke recurrence | 48 weeks (second stage)
  Difference in stroke recurrence rate of butylphthalein treatment compared with routine stroke treatment at 48 weeks
Changes of mRS at 48 weeks compared with baseline. | 48 weeks (second stage)
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The mRS is a range from 0-6. 0=No symptoms, 1=No significant disability. Able to carry out all usual activities, despite some symptoms. 2=Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3=Moderate disability. Requires some help, but able to walk unassisted. 4=Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5=Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6=Dead

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Incidence of Treatment-Emergent Adverse Events [Safety]
Dropout rates and reasons [Safety] | 12 weeks, 24 weeks, 36 weeks and 48 weekss
  Dropout rates and reasons [Safety]

CONTACTS AND LOCATIONS:
Locations (1):
- Donggang Center Hospitol, Dandong, Liaoning, China